CLINICAL TRIAL: NCT05996081
Title: A Practical Adherence Toolkit for Managing Nonadherence to HIV Medications in Indonesia: Protocol for a Usability Study and Cluster Randomised Controlled Trial
Brief Title: Adherence Toolkit for Managing Nonadherence to HIV Medications in Indonesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Groningen (Other)
Collaborators: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Zamrotul Izzah, PhD candidate, University of Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: V1-072023
Record Dates: First submitted 2023-07-21; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Adult; HIV Infections
Keywords: Adherence; Antiretroviral therapy; HIV; Medication beliefs; Quality of life; Treatment knowledge
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: A cluster randomised controlled trial consists of two parallel groups: group 1 gets a usual care (control), and group 2 receives a usual care and an adherence toolkit (intervention). The unit of randomisation is HIV clinic. Each HIV clinic will be randomly allocated to the intervention or control group. People living with HIV who are attending the clinic and receiving ART will be screened for their adherence prior to trial initiation. Those who are suspected to be nonadherent to HIV medications will be recruited to participate in the trial. The intervention period will last for 12 months for each participant in the intervention group, with equivalent follow-up period for participants in the control group. Outcome measures will be collected at 0, 3, 6, and 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Individuals in the HIV clinics randomised to the control or intervention group will attend a consultation session as a usual HIV care based on the Indonesian guideline for HIV care and treatment (Ministry of Health Regulation No. 23/2022). Although it may slightly vary by clinic, for every visit they will collect their medications and receive general information from the HIV care provider on the prescribed ART regimens, including the dose, time of administration, potential side effects and how to deal with them, and the importance of adherence. They will be followed-up at the same time points as those in the intervention group.
- Intervention (Experimental): Individuals attending the HIV clinics that are randomised to the intervention group will receive an intervention over 12 months in addition to usual care. The intervention using an adherence toolkit will be delivered during regular clinic visits when they collect their medications.
  Interventions: Behavioral: Adherence toolkit

INTERVENTIONS:
Behavioral: Adherence toolkit — The adherence toolkit consists of a flowchart of adherence intervention, a self-reported adherence questionnaire, and an intervention wheel as a decision support tool for a healthcare provider. The toolkit can guide HIV care providers to identify problems causing nonadherence and to tailor the effective interventions based on the individual problems. It is available in a Bahasa Indonesia version, accompanied by a user guide on the practical application of the intervention, and can be used digitally or printed on paper. The intervention wheel is an integrated HIV medication adherence influencing factors and effective adherence-promoting interventions derived from systematic reviews and meta analyses, including previous studies conducted in Indonesia.
  Arms: Intervention

SUMMARY:
The goal of this usability study and a cluster randomised controlled trial is to investigate the effectiveness of an adherence toolkit as a decision support tool to improve adherence to antiretroviral therapy. The main questions it aims to answer are: 1) is the adherence toolkit useable and acceptable among HIV care providers in Indonesian clinical practice? and 2) is the adherence toolkit superior than the usual care in improving adherence to antiretroviral therapy among people living with HIV in Indonesia? HIV clinics in Surabaya, Indonesia, will be recruited to participate in the study. HIV care providers will be included in the usability study, whereas people living with HIV will be enrolled in the cluster randomised controlled trial. People living with HIV will be randomly assigned in a 1:1 ratio to the control group receiving usual HIV care and the intervention group receiving an intervention using the adherence toolkit in addition to usual HIV care.

DETAILED DESCRIPTION:
Consistent adherence to antiretroviral therapy (ART) is important to maintain viral suppression and good quality of life among people living with HIV. However, maintaining a high level of ART adherence is challenging because adherence is a complex behaviour and many factors contribute to nonadherence. Therefore, a decision support tool is proposed to help HIV care providers in addressing the barriers and providing the adherence-promoting interventions tailored to the individual needs. The present study comprises a usability assessment followed by a cluster randomised controlled trial to investigate the effectiveness of the adherence toolkit as a decision support tool on improving adherence to ART. Twelve HIV clinics in Surabaya, Indonesia, will be randomised 1:1 to the control (usual care) and intervention (adherence toolkit and usual care) group. The intervention period will last for 12 months, with outcome measures will be collected at initiation, 3-, 6-, and 12-month post-initiation. The primary outcome is adherence to ART measured using a self-reported adherence questionnaire and pharmacy refill records. The secondary outcomes include clinical outcomes (viral load, CD4), HIV treatment knowledge, medication beliefs, and health-related quality of life. The findings will enable HIV care providers, people living with HIV, and policy makers to make informed decision about the value of the adherence toolkit for being used in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Doctors, nurses, and pharmacists who have been trained to provide HIV care and treatment by the Indonesian Ministry of Health
* People living with HIV who have been receiving any ART regimens for at least six months, aged 18 years and older, with any coinfection or comorbidity, suspected to be nonadherent to HIV medications (e.g., having sustained treatment interruptions, inconsistent prescription refill, increased viral load >1,000 copies/ml, decreased CD4 count <200 cells/mm3, or developed opportunistic infections), and provided informed consent

Exclusion Criteria:

* People who have severe mental or physical constraints, drop-out or withdraw after the commencement of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to antiretroviral therapy (ART) | 0, 3, 6, and 12 months
  The primary outcome of the trial is the difference in the changes of adherence rates between the intervention and the control group. The outcome will be repeatedly measured as proportion of people who adhere to ART in the intervention and control groups at study initiation and during the follow-up periods using a previously validated self-reported adherence questionnaire and pharmacy refill data.

SECONDARY OUTCOMES:
Viral load | 0 and 12 months
  The viral load test will measure the number of HIV copies in a milliliter of plasma (in copies/ml).
CD4 cell count | 0 and 12 months
  The CD4 cell count will measure the number of CD4 cells in plasma (in cells/mm^3).
HIV treatment knowledge | 0, 3, 6, and 12 months
  HIV treatment knowledge will be assessed using a validated Bahasa Indonesia version of 8-item brief estimate of health knowledge and action-HIV questionnaire. The questionnaire comprises eight statements, three items assessing HIV knowledge and five items evaluating treatment action. Each response is assigned a score of 0, indicating an incorrect, unsure, or disagree answer, or score 1, indicating a correct or agree answer. The total scores range from 0 to 8, and higher scores correspond with adequate HIV treatment knowledge.
Medication beliefs | 0, 3, 6, and 12 months
  Medication beliefs will be examined by a validated Bahasa Indonesia version of the 18-item beliefs about medicines questionnaire. The questionnaire consists of two sections with 18 statements. The general section contains two four-item scales asking about medication beliefs in general, relating to medication harm (General-Harm) and overuse (General-Overuse). The specific section comprises two five-item scales asking about the necessity of prescribed medication (Specific-Necessity) and concerns about its negative effects (Specific-Concerns). The response for each statement is given on a 5-point Likert scale, where 1 means "Strongly disagree" and 5 means "Strongly agree". The total scores for the harm and overuse scales range from 5 to 20, while for necessity and concerns range from 5 to 25. Higher scores denote stronger medication beliefs.
Health-related quality of life | 0, 3, 6, and 12 months
  Health-related quality of life will be determined by a validated Bahasa Indonesia version of the 31-item World Health Organization (WHO) quality of life-HIV brief questionnaire. The questionnaire contains 31 questions that examine general quality of life (questions 1 and 2) and six domains of health-related quality of life including physical health (questions 3, 4, 14, and 21), psychological health (questions 6, 11, 15, 24, and 31), level of independence (questions 5, 20, 22, and 23), social relationships (questions 17, 25, 26, and 27), environmental health (questions 12, 13, 16, 18, 19, 28, 29, and 30), and spirituality/personal beliefs (questions 7, 8, 9, and 10). Individual items are rated on a 5-point Likert scale where 1 indicates a negative perception and 5 indicates a positive perception. Scoring and coding of each domain follows the instructions provided by WHO, so that each domain scores range between 4 and 20 with higher scores reflect better quality of life.
Usability | 1 month
  A Bahasa Indonesia version of validated system usability scale questionnaire will be used to measure the usability of the adherence toolkit. The questionnaire consists of ten statements with answers given on a 5-point Likert scale, ranging from "Strongly disagree" (1) to "Strongly agree" (5). The total scores range from 0 to 100, with a higher score indicating higher perceived usability and a score of 68 is considered the average.
Acceptability | 12 months
  A one-on-one interview will be performed to explore the perception of HIV care providers on acceptance, experience, and room for improvement of the adherence toolkit.

CONTACTS AND LOCATIONS:
Overall Officials: Zamrotul Izzah, MSc, Principal Investigator — Universitas Airlangga
Locations (1):
- HIV clinics, Surabaya, Indonesia

IPD SHARING:
Plan to Share IPD: No
De-identified data will be available only to authorised persons for analysis and reporting purposes.